CLINICAL TRIAL: NCT02720757
Title: Assessment of Physical Functioning and Handling of Spiolto® Respimat® in Patients With Chronic Obstructive Pulmonary Disease (COPD) Requiring Long-acting Dual Bronchodilation in Routine Clinical Practice
Brief Title: Assessment of Physical Functioning and Handling of Spiolto Respimat in Patients With COPD (OTIVACTO)
Status: Terminated | Type: Observational
Why Stopped: Recruitment failure
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.45
Record Dates: First submitted 2016-03-03; First posted 2016-03-28 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Spiolto Respimat: COPD patients requiring a fixed combination therapy of two long-acting bronchodilators (LAMA + LABA) according to approved Summary of Product Characteristics (SmPC) and Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
  Interventions: Drug: Spiolto Respimat

INTERVENTIONS:
Drug: Spiolto Respimat — Tiotropium bromide + Olodaterol

SUMMARY:
The primary objective of this Non Interventional Study is to measure changes in physical functioning, a surrogate for physical activity and exercise capacity, in COPD patients on treatment with Spiolto® Respimat® in routine daily treatment after approximately 6 weeks.

A secondary objective is to evaluate the patient's general condition (physician's evaluation) from Visit 1 (baseline visit at the start of the study) to Visit 2 (final visit at the end of the study, approx. 6 weeks after Visit 1), as well as patient satisfaction with Spiolto® Respimat® at Visit 2.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent prior to participation
2. Female and male patients = 40 years of age
3. Patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD) and requiring long-acting dual bronchodilation (LAMA + LABA) treatment according to approved Spiolto® Respimat® SmPC and COPD GOLD guideline recommendation

Exclusion criteria:

1. Patients with contraindications according to Spiolto® Respimat® SmPC
2. Patients who have been treated with a Long-acting beta2 adrenoceptor agonist\Long-acting muscarinic antagonist (LABA/LAMA) combination (free and fixed dose) in the previous 6 weeks.
3. Patients continuing Long-acting beta2 adrenoceptor agonist Inhalative Corticosteroids (LABA-iCS) treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
5. Pregnancy and lactation
6. Patients currently listed for lung transplantation
7. Current participation in any clinical trial or any other non-interventional study of a drug or device Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD) patients
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- Multiple Locations, Belgium
- Multiple Locations, Denmark
- Multiple Locations, Luxembourg
- Multiple Locations, Netherlands
- One Or Multiple Investigational Sites, Portugal
- One Or Multiple Investigational Site, Sweden

REFERENCES:
- [Derived] Spielmanns M, Tamm M, Schildge S, Valipour A. Swiss Experience in Therapy With Dual Bronchodilation in Chronic Obstructive Pulmonary Disease in Relation to Self-Reported Physical Functionality. J Clin Med Res. 2021 Jul;13(7):392-402. doi: 10.14740/jocmr4542. Epub 2021 Jul 28. PMID 34394782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label observational study conducted in 6 countries, enrolling consented Chronic Obstructive Pulmonary Disorder (COPD) patients who received treatment with Spiolto® Respimat® according to the approved summary of product characteristics (SmPc).
Pre-assignment Details: Patients were enrolled consecutively and were followed over an observational period of approximately 6 weeks, which was the average time between two medical consultations
Groups:
- Tiotropium + Olodaterol FDC: Patients were administered Tiotropium + olodaterol fixed-dose combination (FDC) using the Respimat® inhaler (Spiolto® Respimat® 2.5 microgram/2.5 microgram) as an inhalation solution.
  Tiotropium + olodaterol FDC is an aqueous solution of tiotropium and olodaterol contained in a cartridge. One cartridge is used per inhaler, which is inserted into the device prior to first use
Period: Overall Study
Arm/Group | Tiotropium + Olodaterol FDC
Started | 132
Completed | 114
Not Completed | 18
Not completed — Other reason | 5
Not completed — Loss of contact | 4
Not completed — Informed consent withdrawal | 1
Not completed — Patients wish to withdraw | 2
Not completed — Missing | 3
Not completed — General exclusion | 3

BASELINE CHARACTERISTICS:
Population: Treated set (TS): Patients that were enrolled, registered and received at least one dose of Spiolto® Respimat® were included in the Treated Set.
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.81 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Therapeutic Success After Approximately (Approx.) 6 Weeks After Baseline
Description: "Therapeutic success" is defined as a 10-point increase of physical functioning (PF)-10 between Visit 1 (baseline) and Visit 2 (approx. 6 weeks later) using a PF questionnaire, which is a subdomain of the Short form (SF)-36 patient questionnaire. The PF-10 sub-domain consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little", or "No, not limited at all", with a score of 1, 2, or 3. The scores over the 10 questions will be summed, resulting in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "No, not limited at all"). The final sum of the individual scores will be standardized to a range of 0 to 100 using the following formula: 100*(sum-10)/20.
  Percentage of patients with therapeutic success after approximately 6 weeks after baseline are presented
Time Frame: Visit 1 (baseline) and at Visit 2 (approx. 6 weeks later)
Population: Full analysis set (FAS): Patients that were enrolled, registered and received at least one dose of treatment with Spiolto® Respimat® and had baseline and week 6 visit documented as well as completed all questionnaires were included in FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 107
percentage of participants | 44.90 [32.23 to 54.78]

2. Secondary Outcome: Change in the PF-10 Score From Visit 1 (Baseline) to Visit 2 (Approx. 6 Weeks Later)
Description: Change in PF-10 score was determined by taking into account the individual change of each patient between Visit 1 and Visit 2.
  PF questionnaire, is a sub-domain of the Short form (SF)-36 patient questionnaire. The PF-10 sub-domain consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little", or "No, not limited at all", with a score of 1, 2, or 3. The scores over the 10 questions will be summed, resulting in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "No, not limited at all"). The final sum of the individual scores will be standardized to a range of 0 to 100 using the following formula: 100*(sum-10)/20.
Time Frame: Visit 1 (baseline) and at Visit 2 (approx. 6 weeks later)
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 107
scores on a scale | 7.64 (17.60)

3. Secondary Outcome: General Condition of the Patient Evaluated by the Physician: Physicians' Global Evaluation (PGE)-Score at Visit 1 (Baseline) and at Visit 2 (Approx. 6 Weeks Later)
Description: The treating physician used the Physician's Global Evaluation (PGE) to evaluate the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8(excellent). PGE will be completed before and approx. 6 weeks after treatment initiation.
  Count of patients with PGE score 2, 3, 4, 5, 6, 7, 8 are presented for Visit 1 and Visit 2.
Time Frame: Visit 1 (baseline) and at Visit 2 (approx. 6 weeks later)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 107
Participants
  Visit 1_score (2) | 7
  Visit 2_score (2) | 1
  Visit 1_score (3) | 18
  Visit 2_score (3) | 14
  Visit 1_score (4) | 28
  Visit 2_score (4) | 14
  Visit 1_score (5) | 18
  Visit 2_score (5) | 14
  Visit 1_score (6) | 19
  Visit 2_score (6) | 33
  Visit 1_score (7) | 15
  Visit 2_score (7) | 20
  Visit 1_score (8) | 2
  Visit 2_score (8) | 11

4. Secondary Outcome: Patient Satisfaction With Spiolto® Respimat® - Overall Satisfaction
Description: A patient satisfaction survey is completed at Visit 2, using a 7-point ordinal scale with divisions from very dissatisfied to very satisfied.
  Count of patients with divisions from very dissatisfied to very satisfied are presented.
Time Frame: Visit 2 (approx. 6 weeks post baseline)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 107
Participants
  Very satisfied: 107 | 20
  Satisfied: 107 | 43
  Rather satisfied: 107 | 22
  Neither satisfied nor dissatisfied: 107 | 14
  Rather dissatisfied: 107 | 4
  Dissatisfied: 107 | 3
  Very dissatisfied: 107 | 1

5. Secondary Outcome: Patient Satisfaction With Spiolto® Respimat® - Satisfaction With Inhaling From the Respimat® Device
Description: as for outcome 4
Time Frame: Visit 2 (approx. 6 weeks post baseline)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 107
Participants
  Very satisfied | 25
  Satisfied | 45
  Rather satisfied | 20
  Neither satisfied nor dissatisfied | 10
  Rather dissatisfied | 5
  Dissatisfied | 2

6. Secondary Outcome: Patient Satisfaction With Spiolto® Respimat® - Satisfaction With Handling of the Respimat® Inhalation Device
Description: as for outcome 4
Time Frame: Visit 2 (approx. 6 weeks post baseline)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol FDC
Number analyzed (Participants) | 107
Participants
  Very satisfied | 33
  Satisfied | 45
  Rather satisfied | 14
  Neither satisfied nor dissatisfied | 9
  Rather dissatisfied | 5
  Dissatisfied | 1

ADVERSE EVENTS:
Time Frame: Data to be collected from signing the informed consent onwards until the end of the study; up to 6 weeks
Description: The following had to be collected from signing the informed consent onwards until the end of the study:
  * all Adverse drug reactions (ADRs) (serious and non-serious), related to Spiolto® Respimat®
  * all Adverse Events with fatal outcome (serious adverse events).
  Treated set is the population set used for reporting Adverse events.
Arm/Group | Tiotropium + Olodaterol FDC
All-Cause Mortality (participants affected / at risk) | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

LIMITATIONS AND CAVEATS:
The impact and the interpretation of this non-interventional (NIS) data are limited due to the non-interventional study concept

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02720757/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT02720757/SAP_001.pdf